

# **Ethics Application Form**

| Applicant details | | | | |
|---|---|---|---|---|
| <ul><li>✓ Staff</li><li>☐ Postgrad</li><li>☐ Postgrad</li></ul> | oer of staff, a postgrad<br>uate Research Stude<br>uate Taught Student<br>aduate Student | | tgraduate taught student or an | undergraduate student? |
| Please enter your job title Professor | | | | ¥ |
| T lease effici you | ur job uue | Professor | | |
| Applicant details | 3 | | | |
| First Name | Anna | | | |
| Surname | Whittaker | | | |
| Division | Faculty of Health | Sciences and Sport | | |
| Faculty | | | | |
| Email | a.c.whittaker@stir | .ac.uk | | |
| Type of appli | cation | | | |
| ✓ A new pr | cation involve any of t<br>oject with Human part<br>oject with Animals | | | |
| <ul><li>□ A project</li><li>□ An applic</li></ul> | that has already rece | ived ethical review<br>ent to a Project Licence | | |

13 August 2024

| A =1 =1:4 | Const. for Arms |
|---|---|
| Addit | tional factors |
| | Does the proposed project involve reproducing copyrighted work in published form (other than brief citation)? |
| | environment, or archaeological remains and artefacts? |
| V | None of the above |
| NILIC | Investive or Clinical research |
| инэ | Invasive or Clinical research |
| If you | r project involves NHS patients, staff, data or premises we would recommend using the HRA Decision Tool to determine whether |
| • | Research Ethics Committee approval will be required. |
| Pleas | se indicate those that apply to your study or select none of the above |
| | Paguiros approval by an NUS Pagagrah Ethica Committee (PEC) |
| | Requires approval by an NHS Research Ethics Committee (REC) Requires approval ONLY by NHS Research and Development (R&D) with an IRAS form |
| | Requires approval ONLY by NHS Research and Development (R&D) - no IRAS form is required |
| | Health care settings (in the UK or overseas) |
| | Clinical trial or an investigational medicinal product |
| | Clinical investigation and/or study of a medicinal product |
| | Human tissue samples or other human biological samples |
| | Imaging investigations (MRI, ultrasound) |
| | Physical examinations (blood pressure, pulse, respiratory rate) |
| <u>~</u> | Physical tests (other than EEG, BioPac, fNIRS) |
| | Computer tests where there are potential health consequences (dementia, sleep apnoea, depression tests) |
| <u>~</u> | Filming or photography (as part of a health research study or in a health setting/context) |
| | Sample-taking (urine, blood, hair, muscle biopsy) |
| | Ingestion of substances, fluids or alcohol |
| | Health related questionnaires, surveys or interviews where there is the potential to diagnose new health related conditions. |
| | None of the above |
| - | |
| Proie | ect details |
| Pleas | se enter the short title of your project (max 200 characters) |
| dance | Sing Care evaluation |

Reference #: NICR 2021 3735 3607 Page 2 of 17

| Please enter the full title of your project |
|---|
| danceSing Care evaluation |
| Staff - If you have a Worktribe record for this project please make sure the titles are the same. |
| Please add the Worktribe reference for this project |
| n/a |
| Are there collaborators involved in the study? |
| ✓ Yes □ No You will be asked to add details of your collaborators later in the form. |
| Turadina alataila |
| Funding details |
| Project funder |
| n/a |
| Please enter the type of funding |
| Please Select |
| <u> </u> |
| Project duration |
| Project start date |
| 03/09/2021 |
| Project end date |
| 31/05/2023 |

| f different from the project start and end dates |
|---|
| Expected start of data collection |
| 10/01/2022 |
| Expected end of data collection |
| 30/12/2022 |
| lealth and Safety |
| f the proposed project poses any particular physical risks to the researcher(s) or research participants a risk assessment must be |
| signed off by your supervisor or line manager prior to commencing fieldwork. |
| Has a health and safety risk assessment been successfully completed? |
| □ Yes |
| □ Not applicable |
| ✓ In progress |
| Project description |
| Please provide a summary of your project (~half page, one page maximum) describing the topic, and |
| main objectives, a summary of your proposed methodology (e.g. fieldwork, experimental procedures, surveys, interviews, focus groups, standardised testing, video or audio recording). |
| Торіс |
| danceSing Care is a creative health and wellbeing company that offers the care sector bespoke, on-demand |
| music and movement resources. This offering is likely to have significant health, social and mental wellbeing |
| penefits but to date this is largely anecdotal. DanceSing Care would like to conduct a more rigorous research project to help promote and endorse their current offering. |
| Main aims/objectives |
| The SPARKLE team will work with danceSing Care to develop a mixed methods research project (qualitative and quantitative research) to evaluate the impact of their music and movement provision on the health and |
| wellbeing of older people in care homes. |

#### Methods

The University has a number of pre-approved protocols for common research scenarios. If you will be following one of the University's protocols please indicate which one here.

1. Develop a toolkit of measures – We will create an advisory group (from our existing contacts through Stirling 1000 Elders run by Prof Whittaker, danceSing Care staff, care home employees) to develop, pre-trial and refine appropriate measures for this age group and sector and ensure outcomes of interest to the advisory group as being assessed. Based on our experience, the toolkit is likely to include quantitative measures of desired outcomes (i.e., health, wellbeing, social connectedness, loneliness) and qualitative methods such as open-ended questions delivered by online surveys - but potentially also some physical tests (chair sit to stand, mobility e.g. timed up and go) if we are able to visit the care homes - Covid19 permitting. We will assess measures that can be implemented by older people themselves with minimal input from carers, can be completed over a relatively short time frame. We will also develop a semi-structured interview/focus group schedule for use after the intervention.

ADDED [ Regarding the physical function measures, we would be potentially asking participants to undertake some simple tests of physical function. These are still being decided by the Advisory Group. These might include some or all of walking speed over 4m, timed-up-and-go walking speed (from seated, 3m then back to seated), standing balance tests (ability to balance in different positions for 30s), and number of sit-to-stand transitions you can complete in 30 seconds. All tests would be described to participants before conducting them and conducted by trained researchers. Physical function testing would only be offered to participants whom their care team deem would be safe to take part in this aspect. We will minimise the number of tests to reduce participant burden and participants would be given regular breaks if we are running more than one of these tests and in a session that is more than 30 minutes duration. These tests would be once prior to the danceSing Care programme starting and once again at the end after the programme 12 weeks later and take 30min to an hour. ]

2. Evaluate danceSing Care – We will recruit older people in care homes who are new to the danceSing Care online programme to complete the toolkit at baseline and then at follow-up at 12 weeks. We will determine an appropriate sample size based on measures included in the toolkit, and our previous project experience but as this is a bit like a feasibility study, we will recruit as many older adults as possible at a single site. A sub-sample of participants and care home staff will take part in more in-depth qualitative data collection on barriers and facilitators of the programme through a semi-structured interviews or focus groups, respectively, at the end. We will then conduct statistical and qualitative thematic analysis on the data from the toolkit at baseline and follow-up to examine change over time.

Phase 2: For a more robust design, a control group will be sought which will include another site or a group due to start the program later.

After an initial group have run through the baseline, 12w access to the danceSing Care programme and follow-up design we will recruit further participants from different care home sites and randomise them to intervention or wait-list control. The design will be the same as above, except the wait-list control group will start the 12w access to danceSing Care after the intervention group have completed this.

Please be aware that if your methodology changes during your research, it is your responsibility to submit an amendment to your approved application. See the Information button for further advice.

### **GDPR**

Applicants must confirm that they have read and understood the University's guidance on GDPR and that the necessary steps have been considered to protect the data of your participants.

Review the University's guidance on GDPR

I have read and understood the University's GDPR guidance

| V | Involves children or vulnerable adults |
|---|---|
| | Involves personal data that has been obtained without the knowledge of the data subjects |
| | Processing of bio-metric or genetic data |
| | Large scale processing of criminal convictions or special categories of personal data? |
| | Processing of personal data involving new technologies or novel applications of existing technologies |
| | Combining or matching personal data obtained from multiple sources |
| | Tracking geo-location |
| | Using personal data in a way that could significantly affect or have an impact on an individual |
| | Jeopardising the physical health or safety of individuals |
| | Systematic monitoring of publicly accessible areas |
| | Profiling or automated decision-making on a large scale where significant decisions are made impacting on people |

Please upload your completed Data Protection Impact Assessment (DPIA)

#### Documents

| Туре | Document Name | File Name | Version<br>Date | Version | Size |
|---|---|---|---|---|---|
| Data Protection Impact<br>Assessment | Data Protection Approval Form_completed_danceSing Care | Data Protection Approval Form_completed_danceSing Care.docx | 13/09/2021 | 1 | 94.4<br>KB |

# Participants, recruitment and location

None of the above

Please indicate those that apply to your project

Provide details of your participant population and the number of participants required

Include brief characteristics as well as principal inclusion and exclusion criteria.

Inclusion for online survey: Aged 60+ living in a care home, capacity to consent, deemed capable of taking part in the online danceSing care resources and sit-to-stand/walking speed tests safely. Care homes complete their own risk assessment of patients for all activities)

Inclusion for follow-up interview/focus groups: Aged 60+ living in a care home and took part in the online survey part, capacity to consent. OR care home staff e.g. activities managers involved in setting up residents with the danceSing Care online resources and helping to recruit participants.

Exclusion: unable to consent, unable to read English, unable to safely take part in online light physical and social activity or any testing as assessed by care home staff.

#### Describe how and from where participants will be recruited.

danceSIng Care has recruited care home organisations in Scotland and North of England to take part in this evaluation. They will liase with care home managers and activity coordinators about the most suitable home for the initial phase. Care home staff independently conduct risk assessments for all activities and would use this for each resident to gauge suitability of the danceSing online activities for each person (out-with whether they take part in the research or not).

Then within the home the research team and danceSing Care will liase with staff about potential residents to approach with the information sheet. Care home staff will then distribute the PIS and its simplified poster version to engage initial interest.

We will use the simple poster as well as the PIS with care home staff and discuss with care home staff in a meeting of those who will be engaged in recruitment about how to talk about the study and answer any questions before they start recruitment. In this meeting we will emphasise the importance of not trying to coerce participation in those who seem reluctant and also underline that non-participants can still take part in the danceSing care activities even if they opt not to take part in the research element of the project.

Interested residents will then be contacted by the researchers via the care team to invite them to agree to take part, and consent and access the online baseline survey. This survey will include the PIS electronic consent form before moving on to the specific measures.

For the foreseable future these activities will be online but from the initial single arm recruitment phase (phase 1) we would like to explore the possibility of utilising PhD students in face to face data collection (Covid19 permitting access to homes) and training local collaborators (peers, care staff) as citizen scientists to undertake a few physical testing measures, e.g., sit-to-stand and walking speed. However, this needs to be explored with the Advisory Group for feasibility before adding this in as measures so is part of the emergent design. We have added details of physical function testing to the PIS.

Phase 2 will recruit in the same way but will be at a different care home, or with residents who have not yet used the danceSing Care resources previously.

#### Describe where the research activities will take place

for example: online, in a classroom, in a sports facility

Online in care homes for the foreseable future for older people for survey (JISC) and interviews (MSTeams)

Online in MSTeams for care home staff focus groups.

Covid-permitting some brief physical function tests (walking speed, sit to stand) in the care home but this remains to be determined with the Advisory group.

### Describe any incentive participants may receive for participation

For applications that will provide Psychology Undergraduate students with research tokens please ensure that your study follows the Undergraduate Student Participation in Research in the Psychology Division Research Tokens Protocol available from the approved protocol section of the website. You should make reference to the protocol in your answer here.

Unlimited access to the danceSing Care online resources for the duration of the project. Some knowledge about how their own walking speed and sit-to-stand performance compares to other older people.

| Does your proposed study involve v | ulnerable groups? |
|---|---|
| ✓ Yes No | |
| Will you be obtaining membership of Disclosure? | f the Protecting Vulnerable Group (PVG) scheme or a |
| <ul><li>✓ Yes</li><li>☐ No</li><li>☐ Existing PVG member</li></ul> | |
| Please provide confirmation or expl<br>Disclosure will be obtained: | ain how Protecting Vulnerable Groups (PVG) scheme, or a |
| without care home staff present will be<br>commencement of project activities if the care home does not envisage that | e directly involved with study participants on their own required to register with the PVG scheme prior to the hey will have any face to face contact alone. Currently this will be required as researchers will not be alone with |
| residents. | |

#### Will you obtain consent from or on behalf of participants? When, where and how?

Remember to include how long you will allow participants to decide whether or not to take part.

ADDED [Capacity to consent will be assessed by residents' usual care team, including care manager/activities coordinator as is usual practice in this setting including in studies we have previously had approved by NHS ethics committees. This involves their in-depth knowledge of the potential participant, their care plan, their current medical diagnoses including dementia, and their medication as well as their assessment of ability to understand the study when it is discussed with them. This is standard in NHS/care settings to rely on the expertise of the health professionals working directly with patients rather than conducting additional screening assessments at this stage (which of course would require consent). Only participants deemed to have capacity to consent will be approached for recruitment. Where this is uncertain, an initial approach to discuss the study will be used to help assess capacity. Only those deemed to have capacity at this stage will be re-approached to confirm recruitment.

Potential participants will have 48hr from initial approach to decide if they are interested in taking part, including time to ask the care staff and/or research team questions about the project. Care staff will then reapproach after 48hr and give access to the online survey to those who are.

The electronic consent form following reiteration of the PIS will be at the start of the online survey.

ADDED [We have also now added an additional opt in/out consent to physical function testing at the end of the survey.

Verbal assent will be checked prior to conducting any physical function tests.]

Similarly, for the sub-group we invite to interviews (older people) or focus groups (care home staff) we will give them 48hr from invitation and reminder via the PIS and consent form emailed through and then care staff will reapproach the older people with the consent form for interviews if they express an interest. Staff will be asked to consent via the consent form and email this back to us if they are interested in taking part in a focus group.

#### How will consent be recorded?

If written consent will not be obtained, justify it here

Online in the survey for older people, for the interviews/focus groups we will email the consent form to the care home for completion and return by participants.

ADDED [ Verbal assent will be rechecked by the researchers before any physical testing sessions or interviews. We have also now added an additional opt in/out consent to physical function testing at the end of the survey and an additional paper consent form for physical function testing alone. ]

#### **Permissions**

| danceSing Ca<br>ADDED [We had formalised the<br>(attached) and | are activities and oun ave discussed CO e Covid risks and moduli follow the care | ur own data collection. VID risk with the Care H itigations into a risk ass | domes operations managessment which has now arding this as well as ex | ger and been approved | | |
|---|---|---|---|---|---|---|
| Ethical impl Describe any e | | d how you will mitiga | ite them | | | |
| about wellbein<br>participants the<br>reinforced and<br>should they we | ng/mental health al<br>nemselves/care hon<br>d we will also suppl | though in our experience<br>the staff. However, the rig<br>y contact information for<br>and we will recommend | upset by some of the su<br>te this is rare and manag<br>ght to withdraw at any tin<br>the PI who is a Health I<br>I that if they are upset by | geable by<br>me will be<br>Psychologist, | | |
| | | - | aused to participants | s and/or third pa | rties | |
| ror example, lando | wners, institutions, cai | No | | | | |
| Methodolog | ies | | | | | |
| Will the propos | sed research inv | olve the deception of | participants? | | | |
| Will the propos | sed research inv | olve concealment or | covert observation? | | | |
| □ Yes | <b>E</b> | No | | | | |
| Is the project of | design emergent | ? e.g. will elements o | of the research be de | eveloped during | he process of the | ne research? |
| ✓ Yes | □ No | | | | | |

13 August 2024

Reference #: NICR 2021 3735 3607 Page 10 of 17

If any additional consent and permission procedures are required please provide details

For example, permissions to conduct field sampling or from local authorities to access schools

Written agreement between danceSing Care, ourselves and the partner care home organisations to run the evaluation project will be sought by danceSing Care in collaboration with the research team prior to initiating recruitment. It is envisaged that visits to interested care homes and online meetings with staff will help to explain and embed the project. Care homes will

#### Provide details of your emergent design

The psychometric tools and specific questions making up the online survey toolkit and the interview/focus group questions will be developed with our advisory panel as the initial part of the study. However, none of these will be diagnostic tools and will likely be similar to those used in our other approved projects (GOALD GUEP 2021 2080 2106, and CSO Covid19 GUEP 905). We have attached a draft list of what the survey is likely to include and a draft example of likely interview/focus group questions. We will be refining this with our Advisory group and ensuring it is not too burdensome.

We will potentially also be asking participants to undertake some simple tests of physical function. These are still being decided by the Advisory Group. These might include some or all of walking speed over 4m, timed-up-and-go walking speed (from seated, 3m then back to seated), standing balance tests (ability to balance in different positions for 30s), and number of sit-to-stand transitions you can complete in 30 seconds. We will minimise the number of tests to reduce participant burden and participants would be given regular breaks if we are running more than one of these tests and in a session that is more than 30 minutes duration. These tests would be once prior to the danceSing Care programme starting and once again at the end after the programme 12 weeks later.

#### Dissemination

How will the results from this study (include feedback to participants) be disseminated?

We will work with the advisory group to produce outputs (including a report) for the participants which will also be used for marketing purposes to promote and roll-out the danceSing Care programme more widely. The full findings will be submitted as a peer reviewed research publication and potential conference posters for wider dissemination to academics and stakeholders which participants can request.

ADDED [Negative or null findings are just as important for danceSing care and for ourselves in terms of informing the development of ongoing and future interventions therefore these will be treated openly and honestly in the same way as any positive data. While danceSing care may be more inclined to tweet particularly about the positive findings from the research and use these in marketing, to avoid biased reporting overall the report provided to danceSing Care to help the development of their services and the associated research article will present ALL findings for their usage. The anonymised data will also be stored and linked to the research article following publication for open access. ]

#### **Data collection methods**

Does the proposed work involved the remote acquisition of data from or about human participants using the internet and its associated technologies?

Yes

□ No

| Please give details | |
|---|---|
| survey will be online twice in older people, a sub-group of participants will be invited for an online interview/focus group - older people will take part in interviews, care staff in focus groups | |
| Does your project involve data from social media? | |
| □ Yes No | |
| Does the proposed work involve collecting or accessing records of, personal or confidentia | information concerning individuals? |
| ✓ Yes □ No | |
| Collection of confidential information | |
| Concentration of confidential information | |
| Describe how the anonymity of participants and the confidentiality of data will be protected this, both through the research and in the dissemination of findings. | and the specific methods to be used for |
| The online survey will be confidential and identifying information (name, DOB) used to match with the follow-up survey will be removed from the downloaded datafile prior to analysis. This information will be stored in a password-protected file on OneDrive by the research team and will not be accessible by anyone else. Data will be stored separately on OneDrive without identifying person information. Semi-structured interview/focus group recordings will be transcribed and transcriptions anonymised prior to data analysis. Original recordings will be destroyed and transcriptions will be stored in password-protected files on OneDrive. | |
| Who will have access to identifiable information? Describe any potential use of the identifia | ble data by others. |
| only the research team and any care staff assisting with measures completion who already know the participants will have access to the raw data including this information. Processed data will be anonymised before revealing findings to danceSing Care. | |
| Indicate if there are any conditions under which privacy or confidentiality cannot be guarar in this research, explain why. | nteed or, if confidentiality is not an issue |
| n/a | |
| Does the proposed work involve the recording of participants through the use of audio visual | I methods? |
| ₹ Yes □ No | |

13 August 2024

Reference #: NICR 2021 3735 3607

| Please give details |
|---|
| Interviews/focus groups will be videorecorded on MSTeams or Zoom depending on the preference of the participants. Software automatically produces a text transcript of the audio portion of the recording which will be cleaned and used as qualitative data for analysis to address project research questions. |
| Will an external contractor be involved e.g. transcription services, interpreters or fieldworkers? |
| □ Yes ▼ No |
| Data analysis |
| Briefly describe the methods of data analysis |
| Descriptive statistics for the sample demographics and baseline questionnaire responses followed by Repeated measures ANOVA on questionnaire ratings/scores from pre-intervention to post |
| Thematic analysis of answers to open-ended questions in the survey and interview/focus group transcriptions. |
| Data storage |
| Briefly describe the methods of data storage |
| All data will be downloaded from the survey host, anonymised by ID and transferred into an |
| SPSS file. A separate list matching ID and contact details for follow-up will be stored separately. All files will be password protected stored in OneDrive accessible only by the research team. |
| Similarly audiovisual files will be transcribed then anonymised and stored in OneDrive. Original recordings will be destroyed. All data will be stored for 10 years. |
| Conflict of interest |
| Does the principal investigator or any other investigator/collaborator have any direct personal involvement (e.g. financial, share-holding, personal relationship etc.) in the organisations sponsoring or funding that research that may give rise to a potential conflict of interest? |
| □ Yes ☑ No |
| Internal collaborators |

13 August 2024

| Please enter details of University of Stirling co-applicants |
|--------------------------------------------------------------|
| First Name |
| Gemma |
| Surname |
| Ryde |
| 1,740 |
| Division |
| Faculty of Health Sciences and Sport |
| Please enter details of University of Stirling co-applicants |
| First Name |
| Jenni |
| Surname |
| Connelly |
| Division |
| Faculty of Health Sciences and Sport |
| Please enter details of University of Stirling co-applicants |
| First Name |
| Len |
| Surname |
| De Nys |
| Division |
| DIVISION |
| Sport |
| Please enter details of University of Stirling co-applicants |
| First Name |
| Esther |
| Surname |
| Ofosu |

| Division | |
|--------------------------------------------------|---|
| Sport | |
| External collaborators | |
| Please add details of any external co-applicants | |
| First Name | |
| Claire | |
| Surname | |
| Hunt | |
| Organisation | |
| danceSing Care | |
| Please add details of any external co-applicants | |
| First Name | |
| Natalie | |
| Surname | ) |
| Surraine | |
| Garry | |
| Organisation | |
| danceSing Care | |
| Documents | |

The University provides a range of template documents. We would strongly recommend that you use the templates that are available on the research ethics and integrity website.

# Please upload your participant information sheet(s)

| Doci | ıme | nte |
|------|-----|-----|

| Туре | Document Name | File Name | Version<br>Date | Version | Size |
|---|---|---|---|---|---|
| Participant information sheet | danceSing Care Participant Information Sheet Online Survey v2 | danceSing Care Participant Information Sheet Online Survey v2.docx | 17/11/2021 | 2 | 81.4<br>KB |
| Participant information sheet | danceSing Care Participant Information Sheet Online Interview v2 | danceSing Care Participant Information Sheet Online Interview v2.docx | 17/11/2021 | 2 | 88.9<br>KB |
| Participant information sheet | danceSing Care Staff Participant Information<br>Sheet Focus Groups v2 | danceSing Care Staff Participant Information<br>Sheet Focus Groups v2.docx | 17/11/2021 | 2 | 88.5<br>KB |

# Please upload your consent sheet(s)

### Documents

| Туре | Document Name | File Name | Version<br>Date | Version | Size |
|---|---|---|---|---|---|
| Consent<br>Form | danceSing Care_Participant_consent_form_int_FG_v2 | danceSing Care_Participant_consent_form_int_FG_v2.docx | 17/11/2021 | 2 | 1.3<br>MB |
| Consent<br>Form | danceSing Care_Participant_consent_form_PhysFunct_v1 | danceSing Care_Participant_consent_form_PhysFunct_v1.docx | 17/11/2021 | 1 | 1.3<br>MB |

# Please upload copies of recruitment material(s)

#### Documents

| Туре | Document Name | File Name | Version<br>Date | Version | Size |
|---|---|---|---|---|---|
| Participant recruitment materials | danceSing Care Evaluation PIS poster v2 | danceSing Care Evaluation PIS poster v2.pptx | 17/11/2021 | 2 | 519.2<br>KB |
| Participant recruitment materials | danceSing Care Evaluation posters A4 staffresidents_v1 | danceSing Care Evaluation posters A4 staffresidents_v1.pptx | 17/11/2021 | 1 | 2.1<br>MB |

## Please attach copies of questionnaire(s), interview or focus group guides

### Documents

| Туре | Document Name | File Name | Version<br>Date | Version | Size |
|---|---|---|---|---|---|
| Interview schedule/topic guide | Interview_Focus Group potential questions | Interview_Focus Group potential questions.docx | 13/09/2021 | 1 | 1.3 MB |
| Interview schedule/topic guide | Sample survey_full_latest<br>draft_v2_17.11.21 | Sample survey_full_latest<br>draft_v2_17.11.21.docx | 17/11/2021 | 2 | 949.1<br>KB |
| Interview schedule/topic guide | danceSing Care physical function tests_draft | danceSing Care physical function tests_draft.docx | 17/11/2021 | 1 | 41.6<br>KB |

# If relevant, please attach copies of debrief information

## If relevant, please attach other documentation

| Docu | 10000 | +- |
|------|-------|----|

| Туре | Document Name | File Name | Version<br>Date | Version | Size |
|---|---|---|---|---|---|
| Other documentation | RA0X-Physical Function-testing-dynamic-and-<br>static | RA0X-Physical Function-testing-dynamic-and-<br>static.docx | 17/11/2021 | 1 | 30.4<br>KB |
| Other documentation | COVID19 risk assessment for fieldwork phys funct testing | COVID19 risk assessment for fieldwork phys funct testing.docx | 17/11/2021 | 1 | 72.9<br>KB |
| Other documentation | Response to Ethics | Response to Ethics.docx | 17/11/2021 | 1 | 25.8<br>KB |

Signing the form will lock the form and prevent further editing. If you choose to unlock the form all signatures will be invalidated and requests will need to be made again.

Please sign your application

Signed: This form was signed by Anna Whittaker (a.c.whittaker@stir.ac.uk) on 19/11/2021 14:12